CLINICAL TRIAL: NCT06957587
Title: Quantitative Estimation of Preoperative Blood Volume Using Multi-modal Ultrasound and Deep Learning
Brief Title: A Deep Learning Model for Blood Volume Estimation From Multi-modal Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng WANG, attending doctor, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-228(K)
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Blood Volume Analysis; Ultrasound; Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients prepare to receive surgery: The patients aged 18-75 years old prepare to receive surgery will be assigned into the cohort.

SUMMARY:
1. Background & Rationale:

   Accurate assessment of a patient's blood volume (BV) status before surgery is critical for preventing perioperative complications. However, there is currently no clinically feasible, accurate, and non-invasive method for direct BV quantification. We hypothesize that dynamic ultrasound videos of major blood vessels contain rich, sub-visual spatiotemporal information about vascular compliance and filling that can be leveraged to estimate BV.
2. Objective:

   To develop and validate a deep learning model that integrates multi-modal ultrasound video data to achieve non-invasive, quantitative estimation of preoperative blood volume.
3. Study Design:

   A prospective, single-center, observational study.
4. Methods:

   Participants: Adult patients scheduled for surgery.

   Data Acquisition:

   Input (Features): Preoperative ultrasound video clips will be recorded in standardized views of four key vessels: the Internal Jugular Vein (IJV), Subclavian Vein (SCV), Inferior Vena Cava (IVC), and Common Carotid Artery (CA).

   Target (Label): The true Blood Volume (BV) will be calculated for each patient using the acute normovolemic hemodilution (ANH) method. The change in hemoglobin concentration before and after this process is used to calculate the total blood volume with high clinical reliability.

   Model Development: A hybrid deep learning architecture (e.g., CNN + LSTM/Transformer) will be trained to extract features from the ultrasound videos and learn the complex, non-linear mapping to the BV value derived from ANH. The model will be trained and internally validated using a k-fold cross-validation approach.
5. Expected Outcome & Significance:

We anticipate the development of a novel, end-to-end deep learning model capable of providing a quantitative BV estimate from routine ultrasound scans. This technology has the potential to revolutionize perioperative fluid management by offering a rapid, non-invasive, and accurate tool for objective volume status assessment, ultimately guiding personalized therapy and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Agree to join this study and sign the informed consent form;
* Age between 18 and 75 years old (inclusive);
* BMI (body mass index) is between 18 and 30 kg/m2;
* American Society of Anesthesiologists (ASA) grades I-II

Exclusion Criteria:

* Preoperative hemoglobin (Hb) <10g/dl
* Cardiac dysfunction (NYHA class III-IV), respiratory dysfunction (ATS class 2-4), history of liver and kidney dysfunction (such as transaminase / albumin / bilirubin abnormalities, hepatitis history, serum creatinine / urea nitrogen rise, etc.), nervous system abnormalities (those who cannot cooperate due to stroke or its sequelae, Alzheimer, etc.);
* The ultrasonic display of inferior vena cava, internal jugular vein, subclavian vein or common carotid artery is extremely poor, venous thrombosis or anatomical abnormalities;
* Multiple injury with chest, abdomen or brain;
* Pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prepare to receive surgery.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative estimation of blood volume | within 30mins before the surgery
  We will estimate the basic blood volume of the patients quantitatively with the Acute Hemodilution technique before the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided